CLINICAL TRIAL: NCT02200965
Title: The National Health Service (NHS) Choice and Information Revolution - Exploring the Utilization of High Quality Clinical Data Governance Processes to Promote Informed Patient Driven Care in a Locally Integrated English Diabetes Health Economy.
Brief Title: Impact of Individualized Structured Information Provision to the Patients, on Diabetes Related Outcomes
Acronym: WICKED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Royal Wolverhampton Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UKCRN-14324
Record Dates: First submitted 2014-07-22; First posted 2014-07-25 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Diabetes; Care Delivery
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Received a letter on 3 occasions (Active Comparator): My Diabetes, My Information, My Plan Document:
  To deliver a structured, understandable, well designed, user friendly, user developed and approved document / letter to all people with diabetes that contains all information about their key care processes in diabetes to promote self-awareness, patient activation and process completion of their own diabetes outcomes.
  This communication (3 mailings per patient (at 0 and 3 and 6 months) will be distributed to the 50% of the whole epidemiological base of people with diabetes (n=>16,000) with the non-interventional group (that will receive the same document once at 3 months) acting as control.
  Interventions: Other: My Diabetes, My Information, My Plan Document
- Received letter on 1 occasion (Active Comparator): My Diabetes, My Information, My Plan Document:
  To deliver a structured, understandable, well designed, user friendly, user developed and approved document / letter to all people with diabetes that contains all information about their key care processes in diabetes to promote self-awareness, patient activation and process completion of their own diabetes outcomes.
  This communication (3 mailings per patient (at 0 and 3 and 6 months) will be distributed to the 50% of the whole epidemiological base of people with diabetes (n=>16,000) with the non-interventional group (that will receive the same document once at 3 months) acting as control.
  Interventions: Other: My Diabetes, My Information, My Plan Document

INTERVENTIONS:
Other: My Diabetes, My Information, My Plan Document — A structured, understandable, well designed, user friendly, user developed and approved letter has been developed and undergone user acceptability testing for this purpose. It succinctly contains all information mapping to core diabetes care processes, is simple and easy to digest and effective in encouraging self-understanding and prompting self-care and empowering informative engagement with services and care providers. The satisfaction of users with the communicating letter both in a developmental pilot phase has been assessed by user group feedback and patient questionnaire.

SUMMARY:
Health professionals usually lead in the management of long term conditions such as Diabetes. In a conventional professionally driven compliance model of care, patients may be placed in a secondary role. National audits show components of systematic diabetes care consistently fail despite several years of heavy expenditure in the service focused Diabetes Quality and Outcome Framework. To what extent is this due to the nature of that process which may not engage patients nor be focused on informed patient centred concerns? The aim of this research is to determine the effectiveness of a healthcare delivery approach in which patients, empowered with structured guidance and specific information about their diabetes, take decisions to get involved in their diabetes care as determined in hard measures of engagement and outcomes. The methodology will be by a whole population cluster randomised controlled study of an intervention the delivery of an individualised diabetes specific structured report, and we will look at its impact on measured key diabetes access and process outcomes. The contention is that the patients, guided in their understanding of empowerment and enablement, equipped with highly person specific risk stratified outcome based information, and informed regarding which actions they may accordingly take, will be enabled to make a significant and impactful contribution in improvement in their own care . This large scale project can deliver on that research question in a tested , efficient and cost effective manner.

DETAILED DESCRIPTION:
Hypothesis & Aim:

The central aim is to determine whether communication of data structured against key diabetes process and outcomes directly to people with diabetes, with an emphasis on enabling, informing and empowering their engagement with service provision will drive improvement in the key parameters of structured diabetes care access, process and outcomes.

Thus we hypothesise that the communicating letter, which is proven to be readable, informative, valuable and desired in user acceptance analysis can be evidenced to drive engagement of users as demonstrated by measures of access and process and that subsequently attainment of access and process permit the achievement of diabetes clinical outcomes.

Project Design

The trial is designed as a prospective cluster randomised controlled trial of an intervention (structured reporting to patients) on key outcomes (as defined below). All patients with diabetes in Wolverhampton will be randomly allocated to receiving 3 mailings at 0, 3 and 6 months (Active Group) or 1 mailing at 3 months (Control Group) of their structured diabetes report (My Diabetes, My Information, My Plan). Using our pan district integrated diabetes information system, data parameters will be observed at 0, 3, 6 and 12 monthly intervals over the 12 months following the delivery of the report.

The objective will be to determine whether the repeated provision of structured, specific and annotated process and outcome information promotes patients to improve their own health care whether by their own actions and /or by seeking support, advice and help and this will be measured using a Process Score and an Outcome Score - emplacing that it is known that surrogate markers for clinical outcomes in diabetes (eg HbA1c) cannot be improved without service Access and completion of process.

The project will run for 2 years - 6 months set up, 1 year active implementation, 6 months analysis, publication, dissemination and closure. Throughout, evidenced effective methodology will be transitioned into standard NHS process.

Project Feasibility:

The Wolverhampton diabetes service is well integrated across primary and secondary care. A centralized pan district register is established. Data linkage between multiple systems is in place, including direct links between the local GP data warehouse (Graphnet) and all specialist / secondary care systems. Data management and governance systems are in place. Data quality is subject to rolling audit and is consistently at >97% accuracy. Effective use of such data has been demonstrated in care pathways - e.g. the diabetes retinal screening programme (national EQA) and the innovative foot care pathway where Wolverhampton amputation rates are amongst the lowest in the country. The local service has a good track record in clinical research. The project has full support of all key NHS groupings including the local Diabetes GP Commissioning Lead (Dr M Sidhu) and the specialist services Clinical Director. All relevant significant others have been engaged in our local Diabetes Implementation Group - including our large local user group (Wolverhampton Action 4 Diabetes) and the regional office of Diabetes UK. We have run a pilot to test the feasibility and effectiveness of our key intervention (structured diabetes information report). This involved consultation with a diverse diabetes user group and conducting a questionnaire survey with 50 patients attending hospital diabetes clinics. Following translation of learning from that pilot into further NHS process, the project is now fully achievable as proposed.

Data Analysis:

Data will be analysed in SPSS for with and between group (paired and unpaired) effects of the individual process and outcome parameters and the summary scores. Thus access process and outcome scores (as defined) will be calculated at baseline and at 3 monthly intervals over 1 year and analysed to determine within and between group effects by 2 way analysis of variance (a group-by-time repeated measures ANOVA) Significance is set at the 5 % level. Professorial level academic statistical advice is available within the local diabetes research group. A power calculation to predict sample size is not warranted since the entire population (not a sample) is to be studied.

ELIGIBILITY:
Inclusion Criteria:

* All People with diabetes aged over 18 registered in local health economy under Wolverhampton City Clinical Commissioning Group.

Exclusion Criteria:

* All People with diabetes aged less than 18 registered in local health economy under Wolverhampton City Clinical Commissioning Group.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17002 (Actual)
Dates: Start 2013-03; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Assessment of change in completion of nine key care processes in diabetes | 12 months
  Completion of nine key care processes; HbA1C, Serum Creatinine, Urine Albumin Creatinine Ratio, Body Mass Index, Serum Cholesterol, Retinal Screening, Foot Screening, Smoking Status and Blood Pressure in people with diabetes are taken as a standard of structured diabetes care delivery. Failure to complete each process over last 15 months (Failed Process Score (FPS)) will be scored as 1. Therefore an individual can have a FPS from 0-9 based on how many parameters were not completed. A change in the FPS score will be compared between the active and control at the end of 12 months period to assess the impact of provision of individualised patient information on the completion of these key care processes that is taken as a marker of Access and Process. This data will be captured in our electronic centralised district diabetes register that captures these nine key care processes and is updated on monthly.

SECONDARY OUTCOMES:
Assessment of change in surrogate markers that define hard outcomes in diabetes | 12 months
  Only with access and completion of process can intervention be made that results in improvement of all associated diabetes care outcome measures - surrogates for hard endpoints e. g. HbA1C, blood pressure, lipid and Coronary Heart Disease (CHD) risk parameters, smoking cessation, renal markers, and eye and foot outcomes emphasising that over this time frame it is not the expectation that hard endpoints (retinopathy, nephropathy, macro vascular outcome and death) will be influenced but that data will be captured and an assessment of change will be made at the end of 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Syed M R Gillani, MRCP, Principal Investigator — The Royal Wolverhampton NHS Trust; Baldev M Singh, MD, Study Director — Royal Wolverhampton NHS Trust
Locations (1):
- Diabetes Centre, New Cross Hospital, Wolverhampton, United Kingdom

REFERENCES:
- [Derived] Gillani SM, Nevill A, Singh BM. Provision of structured diabetes information encourages activation amongst people with diabetes as measured by diabetes care process attainment: the WICKED Project. Diabet Med. 2015 Jul;32(7):865-71. doi: 10.1111/dme.12737. Epub 2015 Apr 11. PMID 25764229